CLINICAL TRIAL: NCT06100978
Title: Patient-reported Outcomes in Status Epilepticus Requiring Intensive Care Unit Management. A Multicenter Longitudinal Cohort Study
Brief Title: Patient-reported Outcome and Patient-reported Experience After Status Epilepticus
Acronym: POSEIDON2
Status: Recruiting | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Jacq Gwenaelle, Investigator Coordinator, Versailles Hospital
Other Study IDs: P22/08 - POSEIDON 2
Record Dates: First submitted 2023-10-15; First posted 2023-10-25 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Patient Reported Outcomes; Patient Satisfaction; Long Term Outcomes; Status Epilepticus; Intensive Care Unit; Burden; Relatives
MeSH Terms: conditions — Patient Satisfaction; Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Status epilepticus (SE) is a common life-threatening neurological emergency in which prolonged or multiple closely spaced seizures can result in long-term impairments. SE remains associated with considerable mortality and morbidity, with little progress over the last three decades. The proportion of patients who die in the hospital is about 20% overall and 40% in patients with refractory SE. Morbidity is more difficult to evaluate, as adverse effects of SE are often difficult to differentiate from those attributed to the cause of SE. Our experience suggests that nearly 50% of patients may experience long-term functional impairments. The precise description of the consequences of these functional impairments and their impact on quality of life after SE requiring intensive care management has been little studied. Indeed, if cognitive, physical and mental impairments are now identified in the populations of patients who required intensive care under the term postresuscitation syndrome (PICS), neuronal lesions consecutive to the SE itselfor to its cause could be responsible for these different functional alterations.

Thus, the following have been described: (i) cognitive disorders in the areas of attention, executive functions and verbal fluency, visual and working memory disorders, but also spatio-temporal disorders; (ii) physical disorders such as the so-called post-resuscitation polyneuromyopathy; and (iii) mental disorders such as anxiety disorders, depressive states or those related to post-traumatic stress.

Assessment and characterization of patient-reported outcomes is essential to complement the holistic assessment of clinically relevant outcomes from the patient's perspective. The POSEIDON study was a cross-sectional collection of PROs and HR-QOL components, and associated with patient functional outcomes, in those who required ICU management for status epilepticus. We propose here to continue the description of potential alterations after a subsequent ME, namely a longitudinal study (POSEIDON 2) which will also include the evaluation of patient-reported experience (PREMS) and the measurement of family burden.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old or older
* Patients previously included in the ICTAL registry (Status Epilepticus cohort NCT03457831)
* Survivors after ICU management for Status Epilepticus More than 3 months and less than 5 years after ICU discharge

Exclusion Criteria:

* Legal guardianship
* Opposition to participate
* Unread and unwritten French language
* Patient not affiliated to a Social Security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the eligibility criteria will be offered participation in the study.
Sampling Method: Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2024-05-25 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
percentage of global impairment of HRQoL | at 3 month and 12 month
  percentage of global impairment of HRQoL defined by one and/or other of the physical and mental impairments (after dichotomization of the SF 36 summary scores compared to the general population) in patients managed in the ICU for or with SE. 36-Item Short Form Survey (SF-36) (HRQoL)-Ranging score[0-100], a high score indicate better health status.

SECONDARY OUTCOMES:
percentage of cognitive impairment in patients managed in the ICU for or with SE | at 3 month and 12 month
  i)The cognitive complaints questionnaire (Questionnaire de Plainte Cognitive (QPC)(Cognition)- a score=3 or more indicate cognitive complaints
percentage of disability in patients managed in the ICU for or with SE | at 3 month and 12 month
  The Glasgow Outcome Scale extended (Handicap)-Ranging score[1-8] a hight score indicate no handicap A score of 5 to 8 on the GOSE indicate a favorable outcome
percentage of physical dependency in patients managed in the ICU for or with SE | at 3 month and 12 month
  The Lawton IADL (scale contains eight items, with a summary score from 0 (low function) to 8 (high function).and Barthel index (Dependency)-Ranging score[0-100], a high score indicate no dependency.
percentage of anxiety and depression in patients managed in the ICU for or with SE | at 3 month and 12 month
  The Hospital anxiety and depression (Anxiety,Depression)-Ranging score[0-21] a score > 8 indicate in each subscale a depresion or/and anxiety
percentage of post traumatic syndrome disorder in patients managed in the ICU for or with SE | at 3 month and 12 month
  The Impact of Event Scale -Revised(post traumatic syndrome disorder)-Ranging score[0-88],scores higher than 24 are of concern; the higher scores indicate the severity of PTSD
score of perceived social support by the SSQ6 scale in its 2 dimensions, satisfaction and availability. | at 3 month and 12 month
  The Social Support Questionnaire- Short Form-SSQ6 / 6 item measure of social support, with scores ranging from 0 (no social support) to 6 (very high social) and 1 (very dissatisfied) to 6 (very satisfied) for the area of satisfaction in each item or area. From these scores in the 6 domains, an average score with the support given in each of the areas.
Presence or absence Post-ICU factors associated of return to work ability in patients managed in the ICU for or with SE. | at 3 month and 12 month
  A return to work will be interpreted by measured by the Work Productivity and Activity Impairment Questionnaire: General Health (WPAI-GH scale)
  The WPAI-GH consists of six questions: 1 = currently employed; 2 = hours missed due to health problems; 3 = hours missed other reasons; 4 = hours actually worked; 5 = degree health affected productivity while working (using a 0 to 10 Visual Analogue Scale (VAS)); 6 = degree health affected productivity in regular unpaid activities (VAS).. Four main outcomes can be generated from the WPAI-GH and expressed in percentages by multiplying the following scores by 100:
patient's experience of the care system. | at 3 month and 12 month
  Score measured by the PPE 15 (Picker Patient Experience Questionnaire) of the patient's experience of the healthcare system.
  It consists of 15 questions distributed to seven dimensions of care: respect, coordination, information/communication/education, physical comfort, emotional support, involvement of relatives, and transitions and continuity The questions have two ("yes" or "no") to four response options ("yes"," no", "I did not need to", or "yes, to some extent"). Neutral answers, such as "I did not need to", and the most positive answer are coded as a "non-problem" (score = 0). The remaining responses are coded as "problems" (score = 1).
experience of the patient's relative at M3 and M12 of discharge from intensive care following management with or for a patient's ME. | at 3 month and 12 month
  Score measured by ZARIT scale Zarit Burden Interview: Revised (22-items) Total score range: 0 to 88 0-21: no to mild burden 21-40: mild to moderate burden 41-60: moderate to severe burden ≥ 61: severe burden

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle Jacq, RN,MSc,PhDc, Study Director — CH Versailles; Stephane Legriel, MD,PhD, Study Director — CH Versailles
Locations (13):
- France (13):
  - CH d'Angoulême, Angoulême
  - CH de Béthune, Béthune
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CH de La Rochelle, La Rochelle
  - CH Versailles, Le Chesnay
  - CHU de Nantes, Nantes
  - Hôpital Paris Saint Joseph, Paris
  - CH de Roanne, Roanne
  - Hôpital Foch, Suresnes
  - CHU Tours, Tours